CLINICAL TRIAL: NCT02055313
Title: The Exceptional Patient in Cancer Care
Brief Title: Perceptions of Exceptional Patients in Cancer Care Relating to Their Unusual Survival
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Moshe Frenkel, Moshe Frenkel MD, Meir Medical Center
Other Study IDs: 2012-1
Record Dates: First submitted 2014-01-30; First posted 2014-02-05 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Cancer; Lung Cancer; Stomach Cancer; Esophageal Cancer
Keywords: Exceptional patient; Cancer care; Lung cancer; Pancreatic cancer; Stomach cancer; Unexplained survival; still alive from 2001-2008
MeSH Terms: conditions — Pancreatic Neoplasms; Lung Neoplasms; Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objective of this study is to explore experiences and insights from exceptional patients, patients with cancer that were considered by their physicians as having exceptional course of survival related to their specific disease state.

A secondary future objective of this study is to develop an international multicenter registry and database documenting and examining the experience of patients with cancer that were considered by their physicians as having exceptional course of survival related to their specific disease state.

DETAILED DESCRIPTION:
This pilot study will utilize a population registry in one location (Israel) to identify exceptional patients with one terminal disease. Pancreatic malignancy, advanced lung cancer; advanced stomach cancer and advanced esophageal cancer have been chosen as the specific terminal disease, based on its extremely high mortality rate. These specific situations can apply to a strict definition set by Gotay: "An exceptional survivor is a cancer patient who is alive when the probability of doing so was less than 25% of living for five or more years , for a given type and stage." [48] These types of cancers are associated with a 5 year survival of less than 15% and even with the latest technology and advances in cancer care; there is a very slight improvement in survival of these patients.

The study will be divided into three stages:

1. Identifying the patients Clalit HMO will be approached to obtain ethical committee's approval to the study and access to the HMO registry. Clalit HMO is the largest HMO in Israel with over 4 million members (out of a total population of 7.5 million). After securing this approval, patients will be identified through the HMO registry. We will try to identify patients with a diagnosis of pancreatic cancer advanced lung cancer, advanced stomach cancer and advanced esophageal cancer that are still alive from 2001-2008.

   Each patient's physician will be contacted to verify that the diagnosis is correct. The physician will be asked to contact the patient and obtain his or her consent to participate in the study. Consenting patients will be sent a letter signed by their primary physician that describes the study and indicates that someone will be calling them to invite them to participate in the study. The letter will clarify that participation is completely voluntary and declining to participate will not affect them in any way.
2. Approaching the patients Patients consenting to participate in the study will be contacted by our qualitative researcher (SG) which will interview them following a qualitative study protocol
3. Analysis of findings and preparation of summary report.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older Ability to speak and read Hebrew, English or Russian. Diagnosis of pancreatic adenocarcinoma advanced lung cancer, advanced stomach cancer and advanced esophageal cancer confirmed by the treating physician, laboratory tests and medical imaging techniques.

Pancreatic adenocarcinoma patient advanced lung cancer, advanced stomach cancer and advanced esophageal cancer patient who is alive when his probability of doing so was less than 15%.

Consent to participate in this study

-

Exclusion Criteria:

* Inability to understand the intent of the study Medical condition that would preclude participation in an interview session lasting over 30 minutes Diagnosis of active psychosis or severe cognitive impairment confirmed by the patient's attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified through the HMO registry in a region of 630,000 members with a diagnosis of pancreatic cancer, advanced lung cancer, advanced stomach cancer and advanced esophageal cancer that are still alive from 2001-2008.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-05; Primary Completion 2020-10 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Qualitative Data Collection: Patients' Experience of Exceptional Disease Course | Two years
  Understanding the patient's experience of a disease process is important in assessing and treating a complicated illness. Qualitative research allows participants to describe an experience in the way that is most meaningful to them. A qualitative approach is deemed as the most appropriate to capture the perceptions and experiences of exceptional patients. This study is using an exploratory, qualitative approach consisting of in-depth, semi-structured interviews. This approach has been widely used in health care to better understand the patient experience. Descriptive analysis of sociodemographic, disease-related, and treatment-related factors were conducted to characterize the sample and to verify that sampling criteria were met. The study endpoint is aimed at reaching saturation of recurring themes that were extracted in the interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe A Frenkel, MD, Principal Investigator — Clalit Health Services

IPD SHARING:
Plan to Share IPD: No